CLINICAL TRIAL: NCT02112305
Title: Comparison Efficacy of Nebulized Magnesium Sulphate to Intravenous Magnesium Sulphate in Children With Severe Acute Asthma
Brief Title: Compare Efficacy Nebulized and Intravenous Magnesium Sulphate in Thai Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Queen Sirikit National Institute of Child Health (Other Government)
Responsible Party: Principal Investigator, Tassalapa Daengsuwan, medical doctor, Queen Sirikit National Institute of Child Health
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EC 104/2557
Record Dates: First submitted 2014-04-04; First posted 2014-04-11 (Estimated); Last update posted 2014-11-18 (Estimated); Status verified 2014-11

CONDITIONS: Acute Severe Asthma
Keywords: Magnesium sulphate nebulized
MeSH Terms: conditions — Status Asthmaticus | interventions — Magnesium Sulfate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- isotonic magnesium sulphate (Experimental): 2.5 ml of isotonic magnesium sulphate (150 mg, 245 mmol/L) on three occasional at 20 minutes interval
  Interventions: Drug: isotonic magnesium sulphate
- 50% magnesium sulphate (Active Comparator): magnesium sulphate 50mg/kg/dose intravenous drip in 20 minutes for one dose
  Interventions: Drug: 50% magnesium sulphate

INTERVENTIONS:
Drug: isotonic magnesium sulphate — 2.5 ml of isotonic magnesium sulphate (150 mg, 245 mmol/L) NB on three occasional at 20 minutes interval
  Other Names: magnesium sulfate
  Arms: isotonic magnesium sulphate
Drug: 50% magnesium sulphate — magnesium sulphate 50mg/kg/dose intravenous drip in 20 minutes for one dose
  Other Names: magnesium sulfate
  Arms: 50% magnesium sulphate

SUMMARY:
The purpose of this study is to determine whether nebulized magnesium sulphate is effective in the treatment of acute severe asthma when comparison with intravenous magnesium sulphate

DETAILED DESCRIPTION:
Intervention: At randomization eligible patients were allocated to receive 2.5ml of isotonic magnesium sulphate (150 mg,245 mmol/L) on three occasional at 20 minutes interval or standard treatment 50 mg/kg intravenous magnesium sulphate. The asthma severity score was record at 0,20,40,60,120,180,240 minutes post randomization. Adverse event were assessed at each assessment point. Patients were followed up until discharge from hospital to collect secondary outcome data.

ELIGIBILITY:
Inclusion Criteria:

* Children age 2-15 years presenting with severe asthma or persistent wheeze without responding to conventional therapy

Exclusion Criteria:

* chronic lung disease
* history of adverse reaction form magnesium sulphate
* life threatening condition

Ages: 2 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2014-01; Primary Completion 2015-05 (Estimated); Study Completion 2015-05 (Estimated)

PRIMARY OUTCOMES:
Asthma severity score | 60 minute

SECONDARY OUTCOMES:
Length of stay in the hospital | within 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Tassalapa Daengsuwan, Pediatrician, Study Director — Queen Sirikit National Institute of Child Health
Locations (1):
- Queen Sirikit National Institute of Child Health, Bangkok, Thailand

REFERENCES:
- [Result] Powell CV, Kolamunnage-Dona R, Lowe J, Boland A, Petrou S, Doull I, Hood K, Williamson PR; MAGNETIC study group. MAGNEsium Trial In Children (MAGNETIC): a randomised, placebo-controlled trial and economic evaluation of nebulised magnesium sulphate in acute severe asthma in children. Health Technol Assess. 2013 Oct;17(45):v-vi, 1-216. doi: 10.3310/hta17450. PMID 24144222